CLINICAL TRIAL: NCT02013947
Title: Randomized Controlled Trial to Analyze the Effects of Moderate Altitude Training on Metabolic Parameters in Voluntary Study Participants With Metabolic Syndrome.
Brief Title: Effects of Moderate Altitude Training on Metabolic Parameters in Voluntary Study Participants With Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Pure Mountain Solda (Other)
Collaborators: Department of internal medicine, Central Hospital Bolzano, South Tyrol, Italy (Unknown); Ospedale Generale Di Zona Silandro (Other)
Responsible Party: Principal Investigator, Dr. Gutwenger Ivana, Dr. med. Gutwenger Ivana, Pure Mountain Solda
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: ESF 2/308/2010
Record Dates: First submitted 2013-11-06; First posted 2013-12-17 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Metabolic Syndrome
Keywords: Exercise, moderate altitude, hypoxia, metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity; Hypoxia | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moderate altitude group (Other): 2 weeks of exercise at 1900 meters sea level
  Interventions: Other: 2 weeks of exercise in low and moderate altitude
- low altitude group (Other): 2 weeks of exercise at 400 meters sea level
  Interventions: Other: 2 weeks of exercise in low and moderate altitude

INTERVENTIONS:
Other: 2 weeks of exercise in low and moderate altitude — Group A will spend 2 weeks at an altitude of 1900m and participants absolve a training program (3h, 4x a week, total training time 24h, training intensity 55-65% of maximal heart rate).
  Group B will spend spend 2 weeks at an altitude of 400m and participants absolve a training program (3h, 4x a week, total training time 24h, training intensity 55-65% of maximal heart rate).

SUMMARY:
The metabolic syndrome is a cluster of metabolic disorders (obesity, hyperglycemia, dyslipidemia and hypertension) and it is a risk factor for the development of type 2 diabetes and atherosclerotic cardiovascular disease. There are several definitions for the metabolic syndrome. The AHA/NHLBI (American Heart association/National Heart Lung Blood Institution)and IDF (International Diabetes Federation)2009 criteria are frequently used to comparing data from studies. Prevention or reduction of obesity and lifestyle modification with physical activity is the main therapeutic goal in patients with metabolic syndrome. Recent studies have shown that exercise in moderate altitude or in moderate hypoxia improved glycemic parameters. The influence of training in moderate altitude on circulating metabolites and hormones in terms of substrate utilization is unclear. The adiponectin seems to play an important role in the homeostasis of adipose tissue and in the pathogenesis of the metabolic syndrome and physical activity seems to have a positive effect on adiponectin concentrations. In this study with randomized controlled pretest-posttest-design we want to investigate the effects of physical activity in moderate hypoxia on biomarkers of metabolic syndrome.

DETAILED DESCRIPTION:
Participate can subjects aged 40-70 years with metabolic syndrome according to the definition of AHA/NHLBI and IDF 2009 after declaring orally and written consent and if they authorize to process personal and sanitary data. The study involve 80 subjects with metabolic syndrome. They will be recruited by general practitioner, elect from the principal investigator and invited to participate in the trial. The 80 participants will be randomized in two groups.

Group A, moderate altitude group, 1900 m, 40 participants Group B, low altitude group, 400m, 40 participants Group A will spend 2 weeks at an altitude of 1900m and participants absolve a training program (3h, 4x a week, total training time 24h, training intensity 55-65% of maximal heart rate).

Group B will spend spend 2 weeks at an altitude of 400m and participants absolve a training program (3h, 4x a week, total training time 24h, training intensity 55-65% of maximal heart rate).

Nutrition does not follow any specific diet plan, both groups receive an equivalent balanced feeding.

Clinical examinations at the beginning and at the end of the study laboratory tests well be documented and compared(fasting plasma glucose, triglycerides, HDL-C, LDL-C, insulin, C-peptid, free fatty acids, adiponectin, leptin, HbA1c, Metabolon cluster, c reactive protein, vit D3). Also BMI, BIA bioimpedance analysis, blood pressure, heart rate, egg, Physical status, exercise test.

ELIGIBILITY:
Inclusion Criteria:

waist circumference in men >102 cm, in women >88cm serum triglycerides >150 mg/dl or drug treatment serum HDL cholesterol < 40 mg/dl in men or <50 mg/dl in women or drug treatment blood pressure >130/95 or drug treatment fasting plasma glucose >100 mg/dl or drug treatment 3 from this 5 criteria -

Exclusion Criteria:

positive anamnesis for myocardial infarction,chronic heart disease, cerebral ischemic occurrences , mental and psychic disorders, not controlled hypertension or hyperglycemia, tumor desease, lung disorders,pregnancy

-

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-11; Primary Completion 2013-11 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
exercise test | examination after 2 weeks of exercise

SECONDARY OUTCOMES:
BMI, BIA, metabolic and cardiorespiratory parameters | examination on baseline and after the 2 weeks

OTHER OUTCOMES:
blood pressure, heart rate | at baseline and after 2 weeks of exercise

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Gutwenger, Principal Investigator — Pure Mountain Solda
Locations (1):
- Gutwenger Ivana, Brixen, Bolzano, Italy

REFERENCES:
- [Derived] Gutwenger I, Hofer G, Gutwenger AK, Sandri M, Wiedermann CJ. Pilot study on the effects of a 2-week hiking vacation at moderate versus low altitude on plasma parameters of carbohydrate and lipid metabolism in patients with metabolic syndrome. BMC Res Notes. 2015 Mar 28;8:103. doi: 10.1186/s13104-015-1066-3. PMID 25885799